CLINICAL TRIAL: NCT06725342
Title: Immune Response Dynamics Predicted by Genomic Patterns in Head and Neck Cancer (HNSCC): a Translational Research Study of the Hellenic Cooperative Oncology Group
Brief Title: HNSCC Immuno-genomics Project
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: ΗΕ5R/18
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Molecular Classification of HNSCC
Keywords: head and neck cancer; genomics; immune-related gene expression
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE tissue blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Combined DNA/RNA sequencing on clinical FFPE material (technically challenging; innovative); immuno-genomics test. — Dual extractions (DNA/RNA) will be carried out from macrodissected thick unstained FFPE sections; samples will be measured for adequate quality / quantity; libraries will be constructed separately with each panel and samples will be sequenced in the same chip in an Ion Torrent Proton System, according to the manufacturer's instructions.
  Sequencing results will be called with the Variant Caller for each panel and submitted for initial analysis and annotation to the Ion Reporter pipeline with each DNA and RNA panel

SUMMARY:
For locally advanced and recurrent / metastatic head & neck squamous cell carcinoma (HNSCC), the is an unmet need for the development of efficient treatment combinations, particularly with immune checkpoint inhibitors. HNSCC have been characterized at the genetic / molecular level concerning characteristics of malignancy and potential clinical actionability ; currently, however, the integration of molecular characteristics of both the malignant cells and the host immune response are considered fundamental for the selection of treatment that best suits these patients .

The primary objective of the NCR-17-12885 project is to classify HNSCC for the selection of optimal therapeutic interventions for the patients, based on genomic characteristics and mutational processes operating in these tumours and on the prevailing activated immune pathways.

DETAILED DESCRIPTION:
Herein we propose the development of a combined genomic and gene expression assay for the comprehensive evaluation of HNSCC for the classification of tumors into (a) those with activated checkpoint molecules and activated T cells, likely to respond to checkpoint inhibition in the case of non-operable disease or recurrent disease without prior treatment; (b) those with inducible checkpoint and T cell response prior to the administration of checkpoint inhibitors; (c) those with activated early inflammatory response that needs to be transformed to cell mediated activation; and (d) those with stable genomes and no immune activation probably necessitating induction of genomic instability and T cell activation.

The test to be developed will provide information on the genomic integrity of the tumor and on a global immune related gene expression profile, both by next generation sequencing

ELIGIBILITY:
Inclusion Criteria:

-Patients with locally advanced squamous cell carcinoma of the head and neck who were treated with concurrent chemoradiotherapy (CCRT) with or without induction chemotherapy (IC) or radical surgery +/- radiotherapy for laryngeal tumors.

Exclusion Criteria:

* Age <18 years old
* Non-squamous cell carcinomas of the head and neck.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced squamous cell carcinoma of the head and neck who were treated with concurrent chemoradiotherapy (CCRT) with or without induction chemotherapy (IC) or radical surgery +/- radiotherapy for laryngeal tumors.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Classification of HNSCC based on their genomic and immune-related gene expression characteristics. | 5 years
  To classify HNSCC for the selection of optimal therapeutic interventions for the patients; classification will be based on present genomic characteristics and mutational processes behind them, and on the prevailing activated immune pathways.

SECONDARY OUTCOMES:
Report on analytical performance of the test | 5 years
  (orthogonal validation with dd-sequencing for genomic variants and comparison of RNA sequencing profiles with the existing Illumina DASL gene expression profiling data
HNSCC classification for comparison with (a) PD-L1 IHC (SP263 assay), and (b) the combined IFNG/PD-L1 mRNA ratio (qRT-PCR) | 5 years
  PD-L1 will be tested by immunohistochemistry and IFNG/PD-L1 mRNA ratio by qRT-PCR
Provision of genomic markers predicting for immune status classes | 10 years
  Provision of genomic markers (DNA) predicting for immune status classes (RNA) and vice versa in HNSCC
One step "immuno-genomics test" | 10 years
  Identification of associations between genomic characteristics and immune response-related gene expression, as well as deaminase or other innate mutagen gene expression. Utillization of existing bioinformatics tools. Predictions will be validated for IFNG and PD-L1 expression, different groups of cell mediated cytotoxicity, early and late inflammatory response gene expression, APOBEC and DNA repair gene expression. The aim is to finally produce a simple genomic test (because knowing the genomic status is currently unavoidable) reliably reflecting the status and potential dynamics of the tumor-host microenvironment.
Reclassification of HNSCC with the "immuno-genomics test" | 10 years
  Molecular classification of HNSCC based on immuno-genomics test
Publication of the results | 10 years
  Publication of results for further expolitation